CLINICAL TRIAL: NCT03827525
Title: Cognitive and Behavioral Therapy of Anxiety in Williams Syndrome
Acronym: WILL-COPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Fondation Jérôme Lejeune (Other); association autour des Williams (Unknown); réseau de santé Maladies Rares (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0375
Record Dates: First submitted 2019-01-29; First posted 2019-02-01 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-01

CONDITIONS: Williams Syndrome; Anxiety
Keywords: Williams Syndrome; Anxiety; Cognitive and Behavioral Therapy; Intellectual Disability
MeSH Terms: conditions — Williams Syndrome; Anxiety Disorders; Intellectual Disability | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Salivary sample will be obtained to evaluate salivary cortisol. Then the sample will be destroyed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cognitive and Behavioral Therapy: There is no group, the study will be based on single case method. The sudy concerns 5 patients with a Williams Syndrome
  Interventions: Behavioral: Cognitive and Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive and Behavioral Therapy — 9 sessions of Cognitive and Behavioral Therapy will be realised with the patient by a clinical psychologist. They will last between 1h and 1h30.

SUMMARY:
Patients with Williams-Beuren syndrome are eight times more likely to suffer from anxiety compared to the general population. Few therapeutic solutions are proposed to these patients. The objective of this research is to validate a cognitive and behavioral therapy anxiety protocol for patients with this syndrome.

DETAILED DESCRIPTION:
Most studies agree that anxiety disorders are more frequent in people with intellectual disabilities that in the general population. Williams syndrome (WS) is a rare disease, associated with an anxiety rate 8 times higher than in the general population. The therapeutic solutions proposed in this population remain limited, in particular concerning approaches without the use of medication. The objective of the study is to evaluate the effectiveness of a program of Cognitive and Behavioral Therapies (CBT) in Williams Syndrome (WS). For this, an ABA-type protocol will be used. It consists of evaluating the effectiveness of an interventional program longitudinally, using a single case type study. Adults patients with WS and suffering from anxiety will be recruited. They will be enrolled in a program consisting in nine sessions of a psychotherapy program targeting anxiety. There will be a pretherapy visit (day 0), nine sessions of psychotherapy (month 0 to month 5) and a visit 3 month after the end of the therapy (at month 8) : the visit of the end of the research (V10). The expected results will be to validate a psychotherapeutic program for patients with WS suffering of anxiety. This program might be extended to other patients with intellectual disability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Williams Syndrome
* Complaint about anxiety
* 18 years old and more
* Score of 7 or more at the CELF-4 (it is a scale assessing the language)
* informed consent signed

Exclusion Criteria:

* Scoring less than 7 at the CELF-4
* Hearing impairment
* Visual impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 5 adults with a Williams Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2019-08-29 (Actual); Primary Completion 2021-04-29 (Estimated); Study Completion 2021-04-29 (Estimated)

PRIMARY OUTCOMES:
Likert anxiety Scale | From day 0 to month 5.
  Repeated evaluation of his anxiety by the patient with the Likert scale. Each day, the patient quantifies his anxiety with the scale with a score from 0 to 9.

SECONDARY OUTCOMES:
Hamilton Anxiety Scale | This score will be obtained at the pre therapy visit (day 0), at the visit of the end of the therapy (month 5), and at the visit of the end of the research (month 8)
  Hamilton anxiety scale will be realised with the patient by a clinical psychologist. It is an evaluation of the anxiety based on 14 questions and observations of the patient. The questions are rated according to the severity of the symptoms: anxious mood, depressed mood, somatic symptoms...Symptoms are evaluated using 5 degrees of severity, from absence of severity to disabling intensity. The overall score ranges from 0 to 60.
Inhibition score | This score will be obtained at the pre therapy visit (day 0), at the visit of the end of the therapy (month 5), and at the visit of the end of the research (month 8)
  the inhibition will be assessed with the Go/no Go test which last 3 minutes.
salivary cortisol | This sample will be obtained at the pretherapy visit (day 0), and at the visit of the end of the research (month 8).
  The sample will be realised by a nurse. The level of cortisol is related to the level of stress.
WHOQOL-BREF score | This score will be obtained at the pre therapy visit (day 0), at the visit of the end of the therapy (month 5), and at the visit of the end of the research (month 8).
  this scale evaluates the quality of life with 26 questions. For each question, the quality of life is evaluated from very low to very high (5 levels). It will be completed by the person of trust.

CONTACTS AND LOCATIONS:
Overall Officials: Natacha LEHMAN, Principal Investigator — Department of Medical Genetics
Locations (1):
- Arnaud de villeneuve Hospital, Montpellier, Hérault, France

REFERENCES:
- [Background] Vereenooghe L, Langdon PE. Psychological therapies for people with intellectual disabilities: a systematic review and meta-analysis. Res Dev Disabil. 2013 Nov;34(11):4085-102. doi: 10.1016/j.ridd.2013.08.030. Epub 2013 Sep 18. PMID 24051363
- [Background] Royston R, Howlin P, Waite J, Oliver C. Anxiety Disorders in Williams Syndrome Contrasted with Intellectual Disability and the General Population: A Systematic Review and Meta-Analysis. J Autism Dev Disord. 2017 Dec;47(12):3765-3777. doi: 10.1007/s10803-016-2909-z. PMID 27696186
- [Background] Unwin G, Tsimopoulou I, Kroese BS, Azmi S. Effectiveness of cognitive behavioural therapy (CBT) programmes for anxiety or depression in adults with intellectual disabilities: A review of the literature. Res Dev Disabil. 2016 Apr-May;51-52:60-75. doi: 10.1016/j.ridd.2015.12.010. Epub 2016 Jan 22. PMID 26803286
- [Derived] Lehman N, Trouillet R, Genevieve D. Evaluation of the Effectiveness of Therapy for Anxiety in Williams Beuren Syndrome Using a Smartphone App: Protocol for a Single-Case Experiment. JMIR Res Protoc. 2023 Apr 3;12:e44393. doi: 10.2196/44393. PMID 37010888